CLINICAL TRIAL: NCT00938925
Title: Effectiveness of Supplementation With Nail Debridement in Ungual Lacquer Treatment in Podiatry Care on Onychomycosis: Pilot Study of Randomized Control Trial
Brief Title: Effectiveness of Podiatry Care on Onychomycosis (EPOCAON)
Acronym: EPOCAON
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funds
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, PhD, University of Malaga
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 03-2009
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2010-03

CONDITIONS: Onychomycosis
Keywords: aggressive debridement; nail lacquer; onychomycosis; podiatry; chiropody; podiatry care
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nail lacquer plus aggressive debridement (Experimental): Nail lacquer plus aggressive debridement: Will be applied abrasion ungual aggressive, this abrasion will be applied in the beginning of the study, week 0 (baseline), the week 12 and the week 24 and he will follow standard treatment with nail lacquer (Odenil 5%) with 2 weekly applications during 36 weeks.
  Interventions: Procedure: Nail lacquer plus aggressive debridement
- nail lacqer alone (Experimental): Nail lacquer alone: Will be applied exclusively standard treatment with nail lacquer during 36 weeks, according to the usual care
  Interventions: Procedure: Nail lacquer alone

INTERVENTIONS:
Procedure: Nail lacquer plus aggressive debridement — Nail lacquer plus aggressive debridement: Will be applied abrasion ungual aggressive, this abrasion will be applied in the beginning of the study, week 0 (baseline), the week 12 and the week 24 and he will follow standard treatment with nail lacquer (Odenil 5%) with 2 weekly applications during 36 weeks.
  Arms: Nail lacquer plus aggressive debridement
Procedure: Nail lacquer alone — Nail lacquer alone: Will be applied exclusively standard treatment with nail lacquer during 36 weeks, according to the usual care
  Arms: nail lacqer alone

SUMMARY:
Onychomycosis occurs in more than 50% of all pathologies unguinal, affecting the health and quality of life of the patient. Although the investigators have a wide therapeutic arsenal, there is still a disparity when carrying out an effective processing.

Hypothesis/Objectives:

To analyze if the use of the podiatric technique of aggressive unguinal abrasion with micrometer sports, in combination with topical treatment with amorolfin 5% in hairspray, significantly increases the effectiveness clinically as well as mycology.

The investigators will analyze the relationship between this intervention and the quality perception of life related to the health of the nails and the foot.

The investigators will Use results for next validation study in Spanish of the questionnaire NailQoL, as well as validation and reliability of the index SCIO and cost study-effectiveness of the processing.

Method:

The investigators will design a randomized control trial. The town will be recruited, informed prior consent will be obtained from patients of 5 Spanish centers of chiropody, with sample size of 313 patients. There will be a screening of 4 weeks to select patients with onychomycosis infections (clinic and mycology both positives); later the patients will be distributed randomly in 2 groups:

* GROUP AM+AU: Will be administered aggressive unguinal abrasion, weeks 0 (baseline), 12 and 24, followed by standard treatment of amorolfin 5%, two weekly applications during 36 weeks.
* GROUP AM: Will be administered exclusively standard treatment of amorolfin 5%, according to common format. The duration will be 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* People of both sexes with ages between 18 and 75 years.
* Having affected at least the nail out of the first toe of a foot.
* Having a confirmed diagnosis of onychomycosis with positive and evidence clinic mycology (KOH and Cultivation) both positive ones.
* The infection should be caused by a fungus dermatology. Will not afford another type of infection because of the possibility of false positives for pollution exogen.

Exclusion Criteria:

* Having received in 6 previous months some local treatment or systemic for the onychomycosis.
* Having dystrophies or alterations ungulates, apart from the ones specific to the onychomycosis, that could to interfere in the interpretation of results.
* Do not have skills for the application and tracking of the topical treatment with the hairspray ungual.
* Allergy to one of the ingredients of the nail lacquer
* Pregnancy or breastfeeding situation acquaintances at the time of recruitment.
* Use of some abrasive or cosmetic product (ej: nail paint) on the treated nail during the tracking of the study.
* Receiving some type of attendance podology or of Pedicure out of the own ones included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
(Potassium hydroxide) KOH and cultivation negative | pre and post intervention and 6 and 12 months of follow up

SECONDARY OUTCOMES:
Clinical improvements of the onychomycosis, valued with SCIO (Scoring Clinical Index for Onychomycosis) | total score, pre and post intervention and 6 and 12 months of follow up
Quality of life perception related the onychomycosis and foot health by nailQoL and foot health state questionnaire (FHSQ) | total score, pre and post intervention and 6 and 12 months of follow up
Quality of life related general health by euroQol 5-D and SF-12 | total score, pre and post intervention and 6 and 12 months of follow up

CONTACTS AND LOCATIONS:
Overall Officials: Irene Garcia-Paya, DPM, MSc, Principal Investigator — University of Malaga; Jose A Sanchez-Castillo, DPM, MSc, Principal Investigator — University of Malaga; Antonio I Cuesta-Vargas, PhD, Study Director — University of Malaga
Locations (3):
- Spain (3):
  - School Health Sciences, University of Malaga, Málaga, Málaga
  - Antonio Cuesta-vargas, Málaga
  - Health Science School , University of Malaga, Málaga

REFERENCES:
- See also: University of Malaga — http://www.uma.es/
- See also: Regional Panel clinicals trials — http://www.juntadeandalucia.es/salud/principal/documentos.asp?pagina=ec_op1
- See also: R+D Spain — http://www.plannacionalidi.es/plan-idi-public/